CLINICAL TRIAL: NCT01684449
Title: Phase 1/2, Randomized, Multicenter, Prospective Study of Gemcitabine and Rapamycin (Sirolimus) Combination Versus Gemcitabine Only to Treat Advanced Soft Tissue Sarcoma
Brief Title: Gemcitabine Plus Rapamycin Versus Gemcitabine to Treat Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-24; 2009-017232-41 (EudraCT Number)
Record Dates: First submitted 2011-06-30; First posted 2012-09-13 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Advanced Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma; Gemcitabine; Rapamycin; Sirolimus; mTOR inhibitor; Molecular biomarkers
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 2: Experimental Arm (Experimental): Gemcitabine + rapamycin at recommended dose of Phase 1. Recommended dose is defined as, the dose one level below of the (MTD). Being MTD, the dose of the cohort in which a maximum of one patient of 6 has presented dose-limiting toxicity (DLT).
  Interventions: Drug: Gemcitabine + Rapamycin

INTERVENTIONS:
Drug: Gemcitabine + Rapamycin — Gemcitabine + rapamycin at recommended dose of Phase 1. Recommended dose is defined as, the dose one level below of the (MTD). Being MTD, the dose of the cohort in which a maximum of one patient of 6 has presented dose-limiting toxicity (DLT).
  Every three weeks until disease progression or unacceptable toxicity. The treatment will last for 6 cycles if there is not progression or intolerable toxicity.
  Additionally, there will be a pharmacokinetic study in a minimum of 9 patients treated with the drug combination.

SUMMARY:
The soft tissue sarcomas (STS) constitute an infrequent group of malignant neoplasms of mesenchymal origin. In Spain, the approximate incidence is of 2 new cases per 100.000 inhabitants every year. In patients with metastatic STS, the average survival is very short, approximately 12 months. The systemic treatment of the metastatic disease has had a very limited development, with few satisfactory results. This facts reflect the urgent need to identify new active agents for treatment of these patients.

The molecular pathway of the serine/threonine kinase mammalian target of rapamycin (mTOR) plays a central role in the regulation of the proteins translation, cellular growth and metabolism (Meric-Bernstam F et al. 2009). Currently, the mTOR pathway is considered a relevant target for the development of anti-cancer drugs, as rapamycin. Preliminary results of some clinical trials suggest that mTOR inhibitors could have some clinical activity for different types of sarcoma, including STS (Chawla et al Proc.ASCO 2006; Schuetze et al. Proc.ASCO 2006).

Gemcitabine is a chemotherapy antimetabolite agent with a broad antitumoral spectrum. The activity of this drug to treat resistant sarcomas and its reduced toxicity make from gemcitabine an adequate candidate for its study in combination with new drugs addressed to molecular targets in the STS treatment.

Pre-clinical studies suggest that mTOR inhibitors could have a potential synergistic or additive effect with some chemotherapy agents. The combination of rapamycin and gemcitabine seems to be a reasonable strategy to explore for the STS treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with anatomopathological diagnosis of metastatic or locally advanced unresectable soft tissue sarcoma (STS). Patients with the following STS types will be excluded: chondrosarcoma, Ewing's sarcoma and embryonal or alveolar rhabdomyosarcoma. In phase 1 it will be allowed to include patients having other types of advanced cancer which are resistant to the standard treatment and can benefit from any of the study drugs.
2. Prior treatment with chemotherapy including doxorubicin and ifosfamide, or contraindication for its administration. The previous treatment with gemcitabine or inhibitors of mTOR is not allowed.
3. Age ≥ 18 y ≤ 70 years.
4. ECOG performance status: 0 - 1. In Phase 1 only patients with ECOG 0-1 will be enrolled.
5. Disease measurable according to RECIST criteria. Proven relapsed disease.
6. Adequate bone marrow function, defined as neutrophil count ≥ 1.500/mm^3 and platelets ≥ 100.000/mm^3.
7. Adequate renal and hepatic function , defined as calculated creatinine clearance ≥ 60 ml/min, creatinine, total bilirubin, AST and/or ALT ≤ 1,5 times the upper limit of normal (ULN).
8. Informed consent form signed by the patient prior to the beginning of the treatment.

Exclusion Criteria:

1. History of previous cancer diagnosed or treated in the past 5 years except basal cell carcinoma, cervical carcinoma in situ or superficial bladder cancer.
2. Presence of brain metastases.
3. Active infection or other severe concomitant diseases.
4. Concurrent treatment with other experimental drugs within 30 days prior to study entry.
5. Pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Phase 1: Determination of dosage: Security and toxicity of the combination gemcitabine and rapamycin. | 15 months
  Type, frequency, seriousness and relation with the treatment of the adverse events in patients treated with the investigational medicinal products.
Phase 2: Progression Free Survival | 12 months
  Progression free survival rate at 3 months to compare the effectiveness of the the treatment.

SECONDARY OUTCOMES:
Phase 2: Overall Survival | 12 months
  Overall survival rate of the patients included in the experimental arm.
Phase 2: Toxicity | 12 months
  Tolerance to the drugs combination of the patients treated with gemcitabine + sirolimus
Phase 1 and 2: Assessment of molecular biomarkers | 36 months
  Assess, both in models of sarcomas induced in immunodeficient mice and tumor samples from patients enrolled in the trial, the predictive value of the response to combination therapy of certain molecular markers for survival and mTOR pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier García del Muro Solans, MD, Study Chair — GEIS
Locations (9):
- Spain (9):
  - H. Sant Pau, Barcelona, Barcelona
  - H. La Paz, Madrid, Madrid
  - H. Son Espases, Mallorca, Mallorca
  - H. Universitario de Canarias, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Instituto Valenciano de Oncología, Valencia, Valencia
  - H. Universitario Miguel Servet, Zaragoza, Zaragoza
  - Institut Català d'Oncologia - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda

REFERENCES:
- [Derived] Martin-Liberal J, Lopez-Pousa A, Martinez-Trufero J, Martin-Broto J, Cubedo R, Lavernia J, Redondo A, Lopez-Martin JA, Mulet-Margalef N, Sanjuan X, Tirado OM, Garcia-Del-Muro X. Phase II Study of Gemcitabine Plus Sirolimus in Previously Treated Patients with Advanced Soft-Tissue Sarcoma: a Spanish Group for Research on Sarcomas (GEIS) Study. Target Oncol. 2018 Feb;13(1):81-87. doi: 10.1007/s11523-017-0539-9. PMID 29177953